CLINICAL TRIAL: NCT05608057
Title: Vitamin C Mesotherapy Versus Diode Laser for the Management of Physiologic Gingival Pigmentation (Randomized Controlled Clinical Trial)
Brief Title: Vitamin C Mesotherapy Versus Diode Laser for the Management of Physiologic Gingival Pigmentation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hams Hamed Abdelrahman (Other)
Responsible Party: Sponsor-Investigator, Hams Hamed Abdelrahman, Assistant lecturer of DPH and Clinical statistician, Alexandria University
Organization: Alexandria University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Laser_VitC2022
Record Dates: First submitted 2022-11-01; First posted 2022-11-08 (Actual); Last update posted 2023-04-27 (Actual); Status verified 2023-04

CONDITIONS: Gingival Pigmentation
MeSH Terms: interventions — Lasers, Semiconductor

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vitamin C mesotherapy (Experimental)
  Interventions: Other: Vitamin C mesotherapy
- Diode laser (Active Comparator)
  Interventions: Radiation: Diode laser

INTERVENTIONS:
Other: Vitamin C mesotherapy — Vitamin C intra-mucosal injection; in which the site of interest will be anesthetized using a topical anesthetic agent (lidocaine gel or xylocaine gel) or infiltration anesthesia, followed by intra-mucosal field injections of 1-1.5 ml Cevarol (L-Ascorbic acid 1000 mg/5 ml
  Arms: Vitamin C mesotherapy
Radiation: Diode laser — Diode laser ablation: in which the site of interest will be anesthetized using infiltration anesthesia, followed by laser ablation. 980nm Diode laser will be applied using the following setting parameters: continuous mode with 980nm wavelength at 1.5 W output power.
  Arms: Diode laser

SUMMARY:
Physiologic pigmentation affects the gingival esthetics. Laser ablation has been recently used as the most effective and reliable technique for gingival depigmentation. However, the high cost of laser technology limits its use in dental practice. Vitamin C/Ascorbic acid mesotherapy has been proposed as a minimally invasive, safe, cost-effective new modality of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Adults between 18 and 45 years old with physiologic melanin pigmentation in the anterior esthetic portion of the maxillary or mandibular gingiva.
* Systemically free

Exclusion Criteria:

* Smokers.
* Drugs intake, which associates with gingival melanin pigmentation.
* Pregnant and lactating women.
* Patients with known hypersensitivity to ascorbic acid.
* Patients with bad oral hygiene.
* Pigmentation of the gingiva due to heavy metal ingestion

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2022-10-22 (Actual); Primary Completion 2023-03-24 (Actual); Study Completion 2023-03-24 (Actual)

PRIMARY OUTCOMES:
Change in gingival pigmentation score | baseline, 1 month, 2 months
  Score 0: Absence of pigmentation Score 1: Spots of brown to black color or pigments. Score 2: Brown to black patches but not diffuse pigmentation Score 3: Diffuse brown to black pigmentation, marginal, and attached gingiva

SECONDARY OUTCOMES:
Change in pain score | up to 1 week
  Visual Analogue Scale (VAS) is a simple measurement tool that measures the intensity of pain as recorded by the patient. 10 point visual analog scale of pain rating, the left side is marked "no pain" and the right side marked "worst pain imaginable.
Patient satisfaction | after 2 months
  After 2 months, patients will be asked to answer three questions to evaluate the level of satisfaction with each technique:
  Did you notice a cosmetic change 2 months after the treatment? (1) No, (2) Moderate, (3) Marked Did treatment meet your expectation? (1) No, (2) yes, (3) Over and above Would you repeat treatment if necessary? (1) No, (2) yes

CONTACTS AND LOCATIONS:
Overall Officials: Sara Esmat, BDS, Principal Investigator — Alexandria University, Faculty of Dentistry
Locations (1):
- Alexandria Faculty of Dentistry, Alexandria, Egypt

REFERENCES:
- [Derived] Esmat SA, El-Sayed NM, Fahmy RA. Vitamin C mesotherapy versus diode laser for the esthetic management of physiologic gingival hyperpigmentation: a randomized clinical trial. BMC Oral Health. 2023 Nov 21;23(1):899. doi: 10.1186/s12903-023-03614-7. PMID 37990224